CLINICAL TRIAL: NCT03367195
Title: Efficacy and Safety of DLBS2411 Compared to Omeprazole in the Management of Gastroesophageal Reflux Disease (GERD)
Brief Title: Efficacy and Safety of DLBS2411 in the Management of GERD
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Very low recruitment rate. The Study Site classifies as tertiary referral hospital. Therefore, GERD Patients being referred to the site are mostly those with comorbidities included in the exclusion criteria.
Sponsor: Dexa Medica Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DLBS2411-0213
Record Dates: First submitted 2017-11-27; First posted 2017-12-08 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Gastroesophageal Reflux Disease (GERD)
Keywords: GERD; DLBS2411; omeprazole
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Omeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment 1 (Active Comparator): 1 Omeprazole capsule 20 mg and 1 placebo caplet of DLBS2411, twice daily
  Interventions: Drug: Omeprazole; Drug: Placebo caplet of DLBS2411
- Treatment II (Experimental): 1 DLBS2411 caplet 250 mg and 1 placebo capsule of Omeprazole, twice daily
  Interventions: Drug: DLBS2411; Drug: Placebo capsule of Omeprazole

INTERVENTIONS:
Drug: Omeprazole — 1 Omeprazole 20 mg capsules twice daily
  Arms: Treatment 1
Drug: DLBS2411 — 1 DLBS2411 caplet 250 mg, twice daily
  Other Names: Redacid
  Arms: Treatment II
Drug: Placebo capsule of Omeprazole — 1 placebo capsule of omeprazole, twice daily
  Arms: Treatment II
Drug: Placebo caplet of DLBS2411 — 1 placebo caplet of DLBS2411, twice daily
  Other Names: Placebo caplet of Redacid
  Arms: Treatment 1

SUMMARY:
This is a 2-arm, prospective, double-blind double-dummy, randomized-controlled study comparing DLBS2411 at a dose of 250 mg twice daily with omeprazole at a dose of 20 mg twice daily, given before morning and evening meals, for an 8-week course of therapy. Subjects should avoid taking meals 2-3 hours before bedtime.

The bioactive fraction of DLBS2411 has been proved at cellular and genetic levels to have an antiulcer effect through both suppressing the gastric acidity and enhancing gastric mucosal protection. The anti-secretory effect of DLBS2411 is exerted through the inhibition of H+/K+ ATPase 'pump' as well as down-regulation of the H+/K+ ATPase gene expression, thus suppressing gastric acid secretion; while its cytoprotective defense mechanism works through the promotion of cyclooxygenase-2 (COX-2) derived prostaglandin (PgE2) synthesis, thus promoting gastrointestinal submucosal blood-flow, stimulating secretion of gastric-epithelial mucous and bicarbonate; anti-oxidative activity; and endothelial-nitric oxide (NO) formation.

Recent study of DLBS2411 which was conducted in healthy volunteers, demonstrated the effective role and safety of DLBS2411 in suppressing intragastric acidity. Having such mechanisms of action, DLBS2411 is hypothesized to benefit patients with gastric acid disorders such as in gastroesophageal reflux disease (GERD).

DETAILED DESCRIPTION:
There will be 2 groups of treatment; each group will consist of 129 subjects with the treatment regimens for 8 weeks:

Treatment I : 1 capsule of Omeprazole 20 mg and 1 placebo caplet of DLBS2411, twice daily Treatment II : 1 caplet of DLBS2411 250 mg and 1 placebo capsule of omeprazole, twice daily

Each study medication will be administered twice daily, 30 minutes before morning (the first) and evening (the last) meals.

The eligible subjects will be randomly allocated to receive study medication (Treatment 1 or Treatment 2) for 8 weeks of treatment, in a double blind fashion. They will be asked to come to the clinic every 4-week interval throughout the study period. Treatment Group 1 will receive Omeprazole twice daily and Placebo DLBS2411 twice daily. While Treatment Group 2 will receive DLBS2411 twice daily and Placebo Omeprazole twice daily.

Subjects will be evaluated for treatment efficacy at baseline and at interval of 4 weeks over the 8-week course of therapy. Throughout the 8-week therapy, subjects should record the frequency (presence and absence) of each of GERD symptoms (heartburn, regurgitation, epigastric pain, nausea) daily in the provided Patient's Diary. The severity of each symptom experienced should also be self-evaluated and recorded.

The safety profile of study medication other than vital signs and adverse event will be measured at baseline and end of study.

Along the study, subjects should avoid taking meals 2-3 hours before bedtime. All subjects will be under direct supervision of a medical doctor during the study period.

ELIGIBILITY:
Inclusion Criteria:

1. Agree to participate in the study under signed informed consent.
2. Male or female subjects aged 18-65 years old.
3. Subjects with diagnosis of GERD confirmed by endoscopy, with esophagitis grade A-B according to the LA Classification.
4. Able to take oral medication.
5. Subjects or subjects' legally acceptable representatives are able and willing to record adverse events in diary.
6. Subjects or subjects' legally acceptable representatives have the ability to comply with the trial protocol, including instruction for taking trial medication.

Exclusion Criteria:

1. For females of childbearing potential: pregnancy and breast-feeding.

   * Patients must accept pregnancy tests during the trial if menstrual cycle is missed
   * Fertile patients must use a reliable and effective contraceptive
2. Subjects with Zollinger Ellison syndrome or peptic ulcer diseases.
3. History or current evidence of Barrett's esophagus, esophageal strictures, odynophagia, pyloric stenosis, esophageal motility disorders (such as achalasia, scleroderma), anatomic esophageal abnormality (such as large hiatal hernia), pill-induced esophagitis.
4. Helicobacter pylori positive as confirmed by urea breath test (UBT).
5. History of esophageal, gastric or intestinal surgery including vagotomy.
6. Presence of comorbid diseases, such as symptomatic coronary artery disease (CAD) or cardiovascular disease, pulmonary disease (including asthma), hemostasis disorder, pancreatitis, malabsorption, or inflammatory bowel disease, and any other chronic diseases (including chronic cough, laryngitis), any serious infection(s), or malignancy(ies).
7. Inadequate liver function defined as ALT or alkaline phosphatase > 2.5 times upper limit of normal.
8. Inadequate renal function defined as estimated Glomerular Filtration Rate (eGFR) < 60 mL/min.
9. Taking any proton pump inhibitors (PPIs) or sucralfate within 14 days prior to screening.
10. Requiring regular and chronic use of non-steroidal anti-inflammatory drugs (NSAIDs), systemic corticosteroids, aspirin, anticholinergics, cholinergics, spasmolytics, or opiates, misoprostol or prokinetics.
11. Hypersensitivity to proton pump inhibitors.
12. Subjects with chronic alcoholism (>40 g alcohol/day) or drug abuse.
13. Active heavy smokers (i.e. consuming >10 cigarettes per day).
14. Participation in any other clinical studies within 30 days prior to screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2020-05-04 (Actual); Study Completion 2020-09-09 (Actual)

PRIMARY OUTCOMES:
Healing rate by endoscopy | 8 weeks
  Healing rate is defined as proportion of subjects with either complete or achieving lower endoscopic grade of esophagitis (according to the Los Angeles (LA) classification) at Week 8 (end of study).

SECONDARY OUTCOMES:
Changes in GERD Questionnaire (GERDQ) sum scores | 4 and 8 weeks
  Changes in GERDQ sum scores from baseline to Week 4 and Week 8 of treatment.
Composite heartburn and regurgitation response rate | 4 and 8 weeks
  Composite heartburn and regurgitation response rate: defined as proportion of subjects with neither heartburn nor acid regurgitation during the last 7 days (complete resolution of heartburn and acid regurgitation) by Week 4 and Week 8.
Heartburn response rate | 4 and 8 weeks
  Heartburn response rate: defined as proportion of subjects with no heartburn during the last 7 days (complete resolution of heartburn) by Week 4 and Week 8 (end of study).
Regurgitation response rate | 4 and 8 weeks
  Regurgitation response rate: defined as proportion of subjects with no regurgitation during the last 7 days (complete resolution of regurgitation) by Week 4 and Week 8 (end of study).
Overall response rate | 4 and 8 weeks
  Overall response rate: defined as proportion of subjects with controlled GERD symptoms by Week 4 and 8 of treatment, defined as proportion categorized as:
  * complete relief (no GERD symptoms during the last 7-day);
  * partial relief (a decrease in frequency but not complete relief of GERD symptoms during the last 7-day); and
  * no response (increase or no change in frequency of GERD symptoms).
Vital sign | 4 and 8 weeks
  Vital sign (blood pressure) from baseline to every follow-up visit including end of study
Electrocardiography (ECG) | 8 weeks
  Electrocardiography (ECG) at baseline and at the end of study
Liver function | 4 and 8 weeks
  Liver function (serum alanine aminotransferase (ALT), serum aspartate aminotransferase (AST), alkaline phosphatase, total bilirubin)from baseline to every follow-up visit including end of study
Renal function | 4 and 8 weeks
  Renal function (serum creatinine and blood urea nitrogen (BUN) level) from baseline to every follow-up visit including end of study
Adverse event | 4 and 8 weeks
  Adverse event, will be observed throughout the study conduct

CONTACTS AND LOCATIONS:
Overall Officials: Dadang Makmun, SpPD, KGEH, Principal Investigator — Division of Gastroenterology Department of Internal Medicine Faculty of Medicine, University of Indonesia Dr. Cipto Mangunkusumo National General Hospital, Jakarta Indonesia; Iswan A. Nusi, Prof. KGEH, FINASIM, FACG, Principal Investigator — Division of Gastroenterohepatology Department of Internal Medicine Faculty of Medicine, University of Airlangga Dr. Soetomo Hospital, Surabaya, Indonesia; Putut Bayupurnama, SpPD, KGEH, Principal Investigator — Division of Gastroenterohepatology Department of Internal Medicine Faculty of Medicine, University of Gadjah Mada Dr. Sardjito Hospital, Yogyakarta, Indonesia; Hery D. Purnomo, SpPD, KGEH, Principal Investigator — Division of Gastroenterohepatology Department of Internal Medicine Faculty of Medicine, University of Diponegoro Dr. Kariadi Hospital, Semarang, Indonesia; Dolvy Girawan, M. Kes., SpPD, KGEH, Principal Investigator — Division of Gastroenterohepatology Department of Internal Medicine Faculty of Medicine, University of Padjajaran Dr. Hasan Sadikin Hospital, Bandung, Indonesia
Locations (5):
- Indonesia (5):
  - Division of Gastroenterohepatology Department of Internal Medicine Faculty of Medicine, University of Padjajaran Dr. Hasan Sadikin Hospital, Bandung
  - Division of Gastroenterology Department of Internal Medicine Faculty of Medicine, University of Indonesia Dr. Cipto Mangunkusumo National General Hospital, Jakarta
  - Division of Gastroenterohepatology Department of Internal Medicine Faculty of Medicine, University of Diponegoro Dr. Kariadi Hospital, Semarang
  - Division of Gastroenterohepatology Department of Internal Medicine Faculty of Medicine, University of Airlangga Dr. Soetomo Hospital, Surabaya
  - Division of Gastroenterohepatology Department of Internal Medicine Faculty of Medicine, University of Gadjah Mada Dr. Sardjito Hospital, Yogyakarta